CLINICAL TRIAL: NCT01777932
Title: A Multicenter, Single-arm, Observational Study Describing the Clinical Benefits of Bevacizumab (Avastin) Treatment in Patients With Metastatic Breast Cancer (AVAREG Study)
Brief Title: AVAREG Study: An Observational Study of Avastin (Bevacizumab) in Patients With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML21647
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Results first posted 2016-02-05 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
This multicenter, single-arm observational study will evaluate the clinical benefits of Avastin (bevacizumab) in combination with paclitaxel in first-line treatment in patients with metastatic breast cancer. Patients with metastatic breast cancer who have started Avastin treatment within 6 months prior to study start will also be eligible. Data will be collected from patients for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic breast cancer initiated on first-line treatment with Avastin in combination with paclitaxel according to the current Hungarian summary of Product Characteristics
* Patients with metastatic breast cancer initiated within 6 months before the start of the study on treatment with Avastin according to the current Hungarian Summary of Product Characteristics

Exclusion Criteria:

Contraindications for Avastin according to the current Hungarian Summary of Product Characteristics:

* Hypersensitivity to active ingredient of Avastin or to any excipients
* Hypersensitivity to products produced in Chinese hamster cells or to other recombinant or humanized antibodies
* Pregnancy
* Untreated central nervous system metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic breast cancer initiated on treatment with Avastin in combination with paclitaxel
Sampling Method: Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2007-12; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Hungary (21):
  - Budapest
  - Debrecen
  - Eger
  - Győr
  - Gyula
  - Kaposvár
  - Kecskemét
  - Kistarcsa
  - Miskolc
  - Nyíregyháza
  - Pécs
  - Salgótarján
  - Szeged
  - Szekszárd
  - Szentes
  - Székesfehérvár
  - Szolnok
  - Szombathely
  - Tatabánya
  - Veszprém
  - Zalaegerszeg

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 220 participants were enrolled across 34 centers in Hungary from 20 December 2007 to 08 March 2011.
Groups:
- Paclitaxel + Bevacizumab Arm: Participants received licensed dose regimens of bevacizumab (10 mg/kg every 2 weeks or 15 mg/kg every 3 weeks) until disease progression, or unacceptable toxicity (whichever occurred first), in accordance with the summary of product characteristics. Paclitaxel could be administered weekly or every 3 weeks according to the accepted oncology protocol.
Period: Overall Study
Arm/Group | Paclitaxel + Bevacizumab Arm
Started | 220
Completed | 15
Not Completed | 205
Not completed — Disease progression | 136
Not completed — Death | 3
Not completed — Adverse Event | 34
Not completed — Lost to Follow-up | 3
Not completed — Investigator decision | 10
Not completed — Reimbursement limit | 9
Not completed — Patient refused further treatment | 10

BASELINE CHARACTERISTICS:
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 187
  >=65 years | 33
Sex/Gender, Customized [Number; unit: participants]
  Female | 218
  Male | 1
  Missing/unknown | 1

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Progression free survival (PFS) was assessed based on time to tumour progression or death (whichever occurred first) from the start of bevacizumab treatment.
Time Frame: Approximately 5 years
Population: All enrolled participants were considered for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
months | 9.3 [7.8 to 10.8]

2. Secondary Outcome: One Year Survival
Description: The status of participants whether alive, dead, unknown or missing one year after the start of bevacizumab treatment is reported.
Time Frame: Approximately 5 years
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
participants
  Alive | 150
  Died | 37
  Unknown | 13
  Missing | 20

3. Secondary Outcome: Time to Discontinuation (TTD) of Bevacizumab Treatment
Description: Time to treatment discontinuation is defined as the time to change of therapy due to any cause (tumour progression, toxicity, or other causes) from the start of bevacizumab treatment.
Time Frame: Approximately 5 years
Population: All enrolled participants were considered for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
months | 7.0 [6.05 to 7.95]

4. Secondary Outcome: Participants With Hormone Receptor Status at Diagnosis
Description: The hormone receptor status for Oestrogen (ER), Progesterone (PgR) and Human epidermal growth factor receptor (HER-2) is reported as positive, negative, unknown or missing.
Time Frame: Baseline (Day 1)
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
participants
  ER positive | 98
  ER negative | 117
  ER unknown | 3
  ER missing | 2
  PgR positive | 90
  PgR negative | 125
  PgR unknown | 3
  PgR missing | 2
  HER-2 positive | 5
  HER-2 negative | 212
  HER-2 unknown | 2
  HER-2 missing | 1

5. Secondary Outcome: Progression Free Survival in Participants With Triple Negative Receptor Status at Study Entry
Description: PFS was assessed based on time to tumour progression or death (whichever occurred first) from the start of bevacizumab treatment for participants with triple negative status and not triple negative status.
Time Frame: Approximately 5 years
Population: All enrolled participants were considered for this outcome measure. Out of the total 220 enrolled participants, 106 participants were triple negative, 110 were not triple negative and data for 4 participants were missing.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
months
  Triple negative (n=106) | 8.30 [7.76 to 8.84]
  Not triple negative (n=110) | 13.30 [10.98 to 15.63]

6. Secondary Outcome: Participants With Tumor Stage at Diagnosis
Description: Number of participants at each Metastatic breast cancer stage 0, I, II, III or IV, at the point of diagnosis is reported.
Time Frame: Baseline (Day 1)
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
participants
  Tumor stage 0 | 1
  Tumor stage I | 38
  Tumor stage II | 87
  Tumor stage III | 39
  Tumor stage IV | 50
  Missing | 5

7. Secondary Outcome: Participants With Eastern Cooperative Oncology Group Status at Study Entry
Description: The Eastern Cooperative Oncology Group (ECOG) status for participants was categorized as 0, 1, 2, or missing. ECOG has 4 grades as: 0 = Fully active, able to carry out all pre-disease activities; 1 = Restricted in strenuous activity but ambulatory and able to carry out work of light or sedentary nature; 2 = Ambulatory and capable of all self-care but unable to carry out work activities. Active about 50% of waking hours; 3 = Capable of limited self-care, confined to bed/chair more than 50% of waking hours; 4 = Completely disabled; cannot carry on self-care, totally confined to bed/chair.
Time Frame: Baseline (Day 1)
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
participants
  ECOG stage 0 | 164
  ECOG stage 1 | 45
  ECOG stage 2 | 7
  Missing | 4

8. Secondary Outcome: Participants With Prior Therapy at Study Entry (Baseline)
Description: The status of prior therapy (i.e. chemotherapy, endocrine therapy, and radiotherapy) at study entry (baseline) is reported.
Time Frame: Baseline (Day 1)
Population: All enrolled participants were considered for this outcome measure
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
participants
  Prior endocrine treatment, Yes | 64
  Prior endocrine treatment, No | 152
  Prior endocrine treatment, Unknown | 1
  Prior endocrine treatment, Missing | 3
  Prior radiotherapy, Yes | 135
  Prior radiotherapy, No | 80
  Prior radiotherapy, Unknown | 2
  Prior radiotherapy, Missing | 3
  Previous chemotherapy, Yes | 127
  Previous chemotherapy, No | 83
  Previous chemotherapy, Unknown | 2
  Previous chemotherapy, Missing | 8

9. Secondary Outcome: Participants With Disease History at Study Entry (Baseline)
Description: Participant's history at the time of diagnosis of metastatic disease and sites of metastases is reported at study entry (baseline).
Time Frame: Baseline (Day 1)
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
participants
  At time of initial diagnosis | 44
  < = 2 years after diagnosis | 91
  > 2 years after diagnosis | 79
  Missing | 6
  Metastatic site, bone | 101
  Metastatic site, lung | 96
  Metastatic site, liver | 65
  Metastatic site, other | 127

10. Secondary Outcome: Participants With Type of Metastases at Study Entry (Baseline)
Description: The type of metastases (bone and visceral) are reported at study entry (baseline) is reported.
Time Frame: Baseline (Day 1)
Population: All enrolled participants were considered for this outcome measure.
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
participants
  Only Bone metastases, Yes | 16
  Only Bone metastases, No | 196
  Only Bone metastases, Missing | 8
  Only Visceral metastases, Yes | 113
  Only Visceral metastases, No | 100
  Only Visceral metastases, Missing | 7

11. Secondary Outcome: Participants With Proteinuria at Study Entry (Baseline)
Description: The number of participants with proteinurea status as positive, negative or missing is reported.
Time Frame: Baseline (Day 1)
Population: All enrolled participants were considered for this outcome measure
Measure: Number; unit: participants
Arm/Group | Paclitaxel + Bevacizumab Arm
Number analyzed (Participants) | 220
participants
  Positive | 3
  Negative | 215
  Missing | 2

ADVERSE EVENTS:
Time Frame: Approximately 5 years
Description: Serious adverse events and non-serious adverse events are reported in all enrolled participants.
Arm/Group | Paclitaxel + Bevacizumab Arm
Serious Adverse Events (participants affected / at risk) | 19/220
Other Adverse Events (participants affected / at risk) | 68/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Bevacizumab Arm (N=220)
Anaemia (Blood and lymphatic system disorders) | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Gastric perforation (Gastrointestinal disorders) | 1
Pain (General disorders) | 1
Acute hepatic failure (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Peritonitis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 2
Blood creatinine increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Nephropathy toxic (Renal and urinary disorders) | 1
Pneumonia (Infections and infestations) | 1
Proteinuria (Renal and urinary disorders) | 3
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2
Embolism venous (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel + Bevacizumab Arm (N=220)
Anaemia (Blood and lymphatic system disorders) | 4
Leucopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 4
Asthenia (General disorders) | 9
Upper respiratory tract infection (Infections and infestations) | 3
Neuropathy peripheral (Nervous system disorders) | 7
Paraesthesia (Nervous system disorders) | 5
Polyneuropathy (Nervous system disorders) | 5
Proteinuria (Renal and urinary disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 4
Nail disorder (Skin and subcutaneous tissue disorders) | 4
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.